CLINICAL TRIAL: NCT04660474
Title: Association of Reperfusion Timing With Short- and Medium-term Ventricular Arrhythmias in Patients With ST-segment Elevation Myocardial Infarction: A Prospective Observational Study
Brief Title: Different Reperfusion Timing and Ventricular Arrhythmias in STEMI Patients
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Affiliated Jiangning Hospital of Nanjing Medical University (Other); The Affiliated Hospital of Hangzhou Normal University (Other); Huai'an First People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VERY-STEMI
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: ST Elevation Myocardial Infarction; Arrhythmia Ventricular
Keywords: Symptom Onset-to-Reperfusion Timing (SO2RT); ST Elevation Myocardial Infarction; Arrhythmia Ventricular; Percutaneous Coronary Intervention; Early Reperfusion
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Early reperfusion group: All patients hospitalized and diagnosed as STEMI according to the 4th universal definition of myocardial infarction underwent coronary angiography and PCI treatment. Patients with SO2RT<24 hours were assigned to Early reperfusion group.
- Intermediate reperfusion group: All patients hospitalized and diagnosed as STEMI according to the 4th universal definition of myocardial infarction underwent coronary angiography and PCI treatment. Patients with SO2RT ranging from 24 hours to 7days were assigned to Intermediate reperfusion group.
- Late reperfusion group: All patients hospitalized and diagnosed as STEMI according to the 4th universal definition of myocardial infarction underwent coronary angiography and PCI treatment. Patients with SO2RT>7days were assigned to Late reperfusion group.

SUMMARY:
The aim of this study was to investigate the association between different reperfusion timing and ventricular arrhythmias (VAs) to provide evidence for clinical decision-making for patients with ST-segment elevation myocardial infarction (STEMI). All the participants included in the study were diagnosed with STEMI according to the 4th universal definition of myocardial infarction, with a follow-up of 1, 6, 12 months, respectively. Symptom onset-to-reperfusion timing (SO2RT) and 24h-dynamic electrocardiogram parameters were recorded to compare different SO2RT and VAs during 3 follow-up visits.

DETAILED DESCRIPTION:
It is Class I recommendation that STEMI require emergency revascularization with no delay. However, arrhythmias after acute myocardial infarction (AMI), particularly VAs, also occur in the early post-MI phase, leading to increased mortality. Previous studies have shown benefits of late reperfusion to electrical stability. The aim of this study was to investigate the association between different reperfusion timing and VAs to provide evidence for clinical decision-making for STEMI. In this multicenter, prospective, observational study, STEMI participants from July 2019 to December 2020 confirmed according to the 4th universal definition of myocardial infarction were enrolled, with a follow-up of 1, 6, 12 months, respectively. SO2RT was defined as the time interval between symptom onset and reperfusion timing which referred to the timing when coronary angiography showed Thrombolysis In Myocardial Infarction (TIMI) blood flow level 2~3 immediately after percutaneous coronary intervention (PCI). The primary end point was VAs on 24h-dynamic electrocardiogram. Secondary outcomes included a composite of death from coronary heart disease, fetal of non-fetal ischemic stroke, revascularization, or chest pain requiring readmission.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients undergoing coronary angiography and PCI;
* can complete 3 follow-up visits well.

Exclusion Criteria:

* without PCI;
* undergoing thrombolytic therapy;
* mental diseases;
* renal failure;
* stroke sequelae;
* tumor and a history of revascularization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective cohort study was designed to investigate the effects of different reperfusion timing on VAs in STEMI patients. During the patients' follow-up, 24h-dynamic electrocardiography, echocardiography were required to record the incidence of primary outcome and other parameters. Information on SO2RT, demographic characteristics, hypertension, diabetes and dyslipidemia history, drug use, smoking, drinking, biochemical indexes and coronary lesions were also collected.
Sampling Method: Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
VAs | 12 months
  The incidence of ventricular arrhythmias on 24h-dynamic electrocardiogram.

SECONDARY OUTCOMES:
Death from coronary heart disease | 12 months
  The incidence of death from coronary heart disease during follow-ups.
Fetal of non-fetal ischemic stroke | 12 months
  The incidence of fetal of non-fetal ischemic stroke during follow-ups.
Revascularization | 12 months
  The incidence of revascularization during follow-ups.
Chest pain requiring readmission | 12 months
  The incidence of chest pain requiring readmission during follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Liansheng Wang, Doctor, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Appleton DL, Abbate A, Biondi-Zoccai GG. Late percutaneous coronary intervention for the totally occluded infarct-related artery: a meta-analysis of the effects on cardiac function and remodeling. Catheter Cardiovasc Interv. 2008 May 1;71(6):772-81. doi: 10.1002/ccd.21468. PMID 18415952
- [Background] Hochman JS, Lamas GA, Buller CE, Dzavik V, Reynolds HR, Abramsky SJ, Forman S, Ruzyllo W, Maggioni AP, White H, Sadowski Z, Carvalho AC, Rankin JM, Renkin JP, Steg PG, Mascette AM, Sopko G, Pfisterer ME, Leor J, Fridrich V, Mark DB, Knatterud GL; Occluded Artery Trial Investigators. Coronary intervention for persistent occlusion after myocardial infarction. N Engl J Med. 2006 Dec 7;355(23):2395-407. doi: 10.1056/NEJMoa066139. Epub 2006 Nov 14. PMID 17105759
- [Background] Malek LA, Silva JC, Bellenger NG, Nicolau JC, Klopotowski M, Spiewak M, Rassi CH, Lewandowski Z, Kruk M, Rochitte CE, Ruzyllo W, Witkowski A. Late percutaneous coronary intervention for an occluded infarct-related artery in patients with preserved infarct zone viability: a pooled analysis of cardiovascular magnetic resonance studies. Cardiol J. 2013;20(5):552-9. doi: 10.5603/CJ.2013.0141. PMID 24297771
- [Background] Sadanandan S, Buller C, Menon V, Dzavik V, Terrin M, Thompson B, Lamas G, Hochman JS. The late open artery hypothesis--a decade later. Am Heart J. 2001 Sep;142(3):411-21. doi: 10.1067/mhj.2001.117774. PMID 11526353
- [Background] Sadanandan S, Hochman JS. Early reperfusion, late reperfusion, and the open artery hypothesis: an overview. Prog Cardiovasc Dis. 2000 May-Jun;42(6):397-404. PMID 10871162
- [Background] Steigen TK, Buller CE, Mancini GB, Jorapur V, Cantor WJ, Rankin JM, Thomas B, Webb JG, Kronsberg SS, Atchison DJ, Lamas GA, Hochman JS, Dzavik V. Myocardial perfusion grade after late infarct artery recanalization is associated with global and regional left ventricular function at one year: analysis from the Total Occlusion Study of Canada-2. Circ Cardiovasc Interv. 2010 Dec;3(6):549-55. doi: 10.1161/CIRCINTERVENTIONS.109.918722. Epub 2010 Nov 9. PMID 21062997